## **Cover page**

**Official Title:** Evaluation of the Communities of HEALing mentorship/support group program:

Assessment of preliminary efficacy

NCT number: NCT03317379

**Document date:** 3/23/2018

## **Statistical Analysis Plan**

Intent-to-treat analyses will be used. Linear mixed models will be used to example the relationship between group (peer, social support, wait list) and each outcome. Predictors in each model will be time, group, and their interaction. For all models, a random intercept will be included. The need for random slopes will be evaluated by examining model fit indices and testing the significance of the difference of the covariance estimate from zero. The peer group will be coded as the reference group to provide estimates and significance values for the difference between peer mentorship and each control condition.